CLINICAL TRIAL: NCT00241189
Title: A 48-week, Double-blind, Randomized, Parallel Phase I/II Study of Oral Rapamycin Versus Methotrexate in Systemic Sclerosis (Scleroderma)
Brief Title: Rapamycin vs Methotrexate in Diffuse SSc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Philip Clements, MD, MPH, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCLA IRB Number: 01-10-045
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Scleroderma; Rapamycin; Methotrexate
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Sirolimus; Methotrexate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapamycin (Experimental): Patients take oral rapamycin 6 mg daily (and dose adjusted to keep a serum trough level of 5-15 ng/ml) for one year
  Interventions: Drug: rapamycin
- Methotrexate (Active Comparator): Methotrexate 20 mg taken orally weekly for one year
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: rapamycin
  Other Names: rapimmune
  Arms: Rapamycin
Drug: methotrexate
  Arms: Methotrexate

SUMMARY:
This is a study to determine the safety of the immunosuppressive rapamycin in patients with systemic sclerosis with diffuse cutaneous scleroderma. The effects (both good and bad) are being compared to another group of systemic sclerosis patients receiving methotrexate

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a disorder characterized by overproduction and deposition of collagen in the skin and visceral organs, abnormalities of the microcirculation, and autoimmunity. Patients who develop extensive skin thickening (diffuse cutaneous scleroderma) usually do so within the first 5 years. In add tion they are at significant risk of early death, severe involvement of heart (10%), lung (15%) and kidney (15-20%) and loss of functional capacity (moderate to severe disability in about 50% within the first few years). there is as yet no proven cure or treatment which prevents heart, lung or kidney damage, prevents disability or improves survival.

In a previsou study, we treated 10 SSc patients with diffuse cutaneous scleroerma with cyclosporin A (CsA), an agent which suppresses the immune response by reducing production of the pro-inflammatory cytokine, interleukin-2 (IL-2). Significant improvement in skin thickening was noted in 6 of the 10 SSc patients. Unfortuantely, significant reduction in kidney function and/or new onset high blood pressure occurred in 8 of the 10. This frequency and degree of adverse events ina population already at risk of kidney failure and high blood pressure is unacceptable.

More recently an immunosuppressive agent with little kidney toxicity, rapamycin, has been found to block the effects of the same pro-inflammatory cytokine as cyclosporin (IL-2) in transplant patients as part of its immunosuppressive action. Since improvement in skin thickening was seen in our patients who received CsA, we postulate that blocking the effects of IL-2 by rapamycin will also result in improvement in skin thickening in SSc patients with extensive skin thickening. There is growing evidence (from our work and the work of others) that softening thick skin in diffuse SSc is associated with improvement in hand function, joint mobility, arthritis signs, overall functional ability, and survival.

The effectiveness of another immunosuppressive, methotrexate, has been compared to placebo (a dummy) in two SSc studies that had a combined total of 100 patients with estensive skin thickening. In both studies there was a trend to greater softening of the thick scleroderma skin. In one study a greater sense of general well being was also noted in the methotrexate group and in the other study the physician global assessment improved to a greater extent in the methotrexate group. Because there is a suggestion of benefit from methotrexate, the present trial evaluating rapamycin is being compared to methotrexte. During a 48 week period rapamycin and methotrexate will be taken as randomly assigned (9 patients in each arm for a total of 18 patients). Over 48 weeks, the status of these patients' scleroderma will be assessed by simple but validated techniques, including simple palpation of the skin to assess skin thickness; lung function texts, electrocardiogram and chest x-ray to assess heart and lungp; blood pressure and serum creatinine to assess kidney; 3 questionnaires (completed by patients) to assess function, quality of life and shortness of breath; and CBC, chemistries and rapamycin levels to assess safety. Statistical analysis of the courses of the two treatment groups will help us determine whether rapamycin has excessive toxicity and whether there are suggestions of efficacy of rapamycin.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy American College of Rheumatology classification criteria for systemic sclerosis
* Have skin thickening proximal to the elbows and/or knees (diffuse scleroderma)
* Cutaneous involvement for less than 5 years from the onset of the first non-Raynaud's manifestation

Exclusion Criteria:

* Severe intractable malabsorption
* Chronic debilitation from any underlying disease
* Off putative disease modifying therapies for one month prior to entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Adverse events
Modified Rodnan Skin thickness score

SECONDARY OUTCOMES:
Forced vital capacity
Diffusing capacity (DLCO)
Health Assessment Questionnaire-Disability Index
Mahler Dyspnea Index
Medical Outcomes Questionnaire SF-36
Patient global (VAS)
Physician global (VAS)
% responders in skin score (=>35% decrease from baseline)
% responders in HAQ-DI(=>0.22 units decrease from baseline)
% responders in FVC (=>10% decrease from baseline)
Serum rapamycin levels

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Clements, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Philip Clements, MD, Los Angeles, California, United States

REFERENCES:
- [Result] Su TI, Khanna D, Furst DE, Danovitch G, Burger C, Maranian P, Clements PJ. Rapamycin versus methotrexate in early diffuse systemic sclerosis: results from a randomized, single-blind pilot study. Arthritis Rheum. 2009 Dec;60(12):3821-30. doi: 10.1002/art.24986. PMID 19950289